CLINICAL TRIAL: NCT00532597
Title: Effects of On-Line Hemodiafiltration(HDF) on Endothelial Dysfunction in Chronic Hemodialysis Patients
Brief Title: Effects of On-Line Hemodiafiltration(HDF) on Vascular Health in Chronic Hemodialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eulji General Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EMCIRB 07-01
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: End Stage Renal Disease; Hemodialysis
Keywords: Vascular Endothelium-Dependent Relaxation; Hemodialysis; Hemodiafiltration
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- O (Experimental)
  Interventions: Procedure: On-line hemodiafiltration
- L (Active Comparator)
  Interventions: Procedure: Low flux hemodialysis

INTERVENTIONS:
Procedure: On-line hemodiafiltration
  Arms: O
Procedure: Low flux hemodialysis
  Arms: L

SUMMARY:
The purpose of this study is to determine whether on-line hemodiafiltration ameliorate the endothelial dysfunction compared with the low flux hemodialysis in end stage renal disease patients on maintenance hemodialysis.

DETAILED DESCRIPTION:
1. On-line hemodiafiltration(OL-HDF) is a technique that combines diffusion with convection in which the large substitution fluid is produced directly from the dialysate. It offers many advantages aside from its safe inflammatory profile, which is attributable to the use of ultrapure dialysate and highly biocompatible dialysis membranes. Due to an improved convective clearance, significantly increased removal of large or protein-bound uremic retention solutes can be achieved, with a potential benefit on cardiovascular morbidity and mortality.
2. Endothelial dysfunction, almost universal in end stage renal disease, is important risk factor for cardiovascular events, and can be evaluated by brachial artery endothelium-dependent vasodilation (flow-mediated dilation) to reactive hyperemia following 5 min of forearm ischemia.
3. The stable HD patients will receive 8-week treatment on OL-HDF or conventional low flux HD and then crossed over to opposite treatment arm. The FMD will be measured by one sonographer, and at the same time whole blood and serum will be sampled and stored for further analysis. The timepoint for measurement is 4-week interval after baseline evaluation.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal disease on maintenance hemodialysis for more than 3 months

Exclusion Criteria:

* diagnosis of active cardiovascular diseases in 6 months
* elevation of liver enzymes over two fold of upper normal limit in 3 months
* admission for acute infection in 3 months
* untreatable stenosis of vascular access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-04; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
endothelial dysfunction measured by flow-mediated vasodilation | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: SuAh Sung, M.D.,PhD., Study Chair — Department of Internal Medicine, College of Medicine, Eulji University
Locations (1):
- Eulji General Hospital, Seoul, South Korea